CLINICAL TRIAL: NCT00511914
Title: A Phase III, Multicenter, Uncontrolled, Open-label Study to Evaluate Safety and Immunogenicity of a Single Intramuscular Dose of a Trivalent Subunit Influenza Vaccine Produced in Mammalian Cell Culture, Using the Strain Composition 2007/2008, When Administered to Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of Trivalent Subunit Influenza Vaccine Produced in Mammalian Cell Culture Using the Strain Composition 2007/2008
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V58P1S; 2007-001404-20
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Results first posted 2013-01-17 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Seasonal Influenza Vaccine
Keywords: Influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cTIV (Adults) (Experimental): Received one dose of cell-culture derived trivalent influenza vaccine (cTIV).
  Interventions: Biological: cTIV
- cTIV (Elderly) (Experimental): Received one dose of cell-culture derived trivalent influenza vaccine (cTIV).
  Interventions: Biological: cTIV

INTERVENTIONS:
Biological: cTIV — One dose (0.5 mL) of cell culture-derived influenza vaccine, administered in the deltoid muscle

SUMMARY:
Annual trial for registration of sub-unit influenza vaccine produced in mammalian cell culture, using the strain composition 2007/2008, when administered to adult and elderly subjects

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrollment into this study are male and female adults who were:

1. ≥ 18 years of age, mentally competent, willing and able to give informed consent prior to study entry
2. available for all the visits scheduled in the study and able to comply with all study requirements
3. in good health as determined by:

   * medical history
   * physical examination
   * clinical judgment of the investigator Written informed consent had to be obtained from all the subjects before enrollment in the study after the nature of the study had been explained.

Exclusion Criteria:

Subjects were not to be enrolled into the study if at least one of the following criteria was fulfilled:

1. Any serious chronic or acute disease such as:

   1. Cancer (leukemia, lymphomas, neoplasm), except for benign or localized skin cancer and non-metastatic prostate cancer not presently treated with chemotherapy
   2. Congestive heart failure
   3. Advanced arteriosclerotic disease
   4. Chronic obstructive pulmonary disease (COPD) requiring oxygen therapy and/or acute exacerbation of a COPD within the last 14 days.
   5. Autoimmune disease (including rheumatoid arthritis), if under immunosuppressive therapy (see below)
   6. Insulin dependent diabetes mellitus
   7. Acute or progressive hepatic disease
   8. Acute or progressive renal disease
   9. Severe neurological or psychiatric disorder
2. History of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study vaccine or chemically related substances
3. Known or suspected (or have a high risk of developing) impairment/alteration of immune function (excluding that normally associated with advanced age) resulting for example from:

   1. Receipt of immunosuppressive therapy (chronic therapy with immunosuppressive drugs, any parenteral or oral corticosteroid (substitution dose in case of absence of suprarenal function allowed) or cancer chemotherapy/radiotherapy) within the last 2 months and for the full length of the study,
   2. Receipt of immunostimulants,
   3. Receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within the past 3 months and for the full length of the study,
   4. Suspected or known HIV infection or HIV-related disease.
4. Known or suspected history of drug or alcohol abuse
5. Bleeding diathesis or receive anticoagulants of the coumarin type
6. Women who are pregnant or woman of childbearing potential unwilling to practice acceptable contraception for the duration of the study (21 days)
7. Influenza immunization or laboratory confirmed influenza within the last 6 months and more than one influenza immunization within the past 12 months
8. Immunization with any other vaccine and/or any investigational vaccine four weeks prior to study start
9. Any significant acute or chronic infections requiring systemic antibiotic treatment or antiviral therapy within the last 7 days
10. Fever (i.e. body temperature ≥ 38.0°C) within the past 3 days prior to study entry
11. Simultaneous participation in another clinical study
12. Any condition, which, in the opinion of the investigator, might prevent the subject from participation or interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2007-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (2):
- Germany (2):
  - Betriebsaerztlicher Dienst, Standort Marburg, Baldingerstrasse, Marburg Hessen
  - Z29, Blutspendezentrale, Gebaude Z29, Behringwerke, Emil-von-Behring-Str. 76, Marburg

RESULTS

PARTICIPANT FLOW:
Groups:
- cTIV (Adults): Adults 18-60 years of age received one dose of cell culture derived trivalent influenza vaccine (cTIV).
- cTIV (Elderly): Elderly subjects >= 61 years of age received one dose of cell culture derived trivalent influenza vaccine (cTIV).
Period: Overall Study
Arm/Group | cTIV (Adults) | cTIV (Elderly)
Started | 68 | 67
Completed | 68 | 67
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | cTIV (Adults) | cTIV (Elderly) | Total
Number analyzed (Participants) | 68 | 67 | 135
Age Continuous [Mean (Standard Deviation); unit: years] | 37.4 (12.3) | 67.4 (4.7) | 52.3 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 25 | 64
  Male | 29 | 42 | 71

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMT) After 1 Dose of Cell Culture Derived Vaccine (cTIV).
Description: Pre and postvaccination geometric mean titers against all 3 strains were assessed by hemagglutination inhibition (HI) assay using egg derived antigen in adults and elderly subjects.
Time Frame: 3 weeks postvaccination (Day 22)
Population: Analysis was done on per protocol set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | cTIV (Adults) | cTIV (Elderly)
Number analyzed (Participants) | 68 | 67
Titer
  A/H1N1 Prevaccination (Day 1) | 22 [14 to 33] | 23 [17 to 31]
  A/H1N1 Postvaccination (Day 22) | 624 [442 to 881] | 199 [150 to 264]
  A/H3N2 Prevaccination (Day 1) | 36 [24 to 56] | 80 [53 to 122]
  A/H3N2 Postvaccination (Day 22) | 405 [299 to 547] | 283 [205 to 390]
  B Prevaccination (Day 1) | 8.16 [6.43 to 10] | 16 [12 to 21]
  B Postvaccination (Day 22) | 96 [66 to 139] | 40 [30 to 53]

2. Secondary Outcome: Number of Subjects Reporting Local and Systemic Reactions
Description: To evaluate the safety and tolerability of cell culture derived vaccine (cTIV) in adults and elderly subjects in terms of number of subjects reporting local and systemic reactions after 1 vaccine dose.
Time Frame: 3 days postvaccination
Population: Analysis was done on safety set.
Measure: Number; unit: Subjects
Arm/Group | cTIV (Adults) | cTIV (Elderly)
Number analyzed (Participants) | 68 | 67
Subjects
  Redness/Erythema | 0 | 2
  Swelling | 2 | 2
  Pain | 31 | 16
  Ecchymosis | 1 | 2
  Induration | 4 | 4
  Fever ( ≥ 38°C) | 0 | 0
  Malaise | 5 | 3
  Fatigue | 10 | 8
  Headache | 12 | 9
  Sweating | 2 | 3
  Myalgia | 3 | 2
  Arthralgia | 4 | 3
  Chills | 0 | 0

3. Primary Outcome: Geometric Mean Ratio After 1 Dose of the Cell Culture Derived Vaccine (cTIV)
Description: Geometric mean ratio (GMR) of Day 22 / Day 1 geometric mean antibody titers was assessed by hemagglutination inhibition (HI)assay using egg derived antigen in adults and elderly subjects.
  The criterion is met according to European (CHMP) guideline if the mean geometric increase GMR (Day22 / Day1) in HI antibody titer is >2.5 for adults and >2.0 for elderly subjects.
Time Frame: 3 weeks postvaccination (Day 22)
Population: Analysis was done on per protocol set
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | cTIV (Adults) | cTIV (Elderly)
Number analyzed (Participants) | 68 | 67
Ratio
  A/H1N1 (Day 22 / Day1) | 29 [18 to 46] | 8.74 [6.13 to 12]
  A/H3N2 (Day 22 / Day1) | 11 [7.27 to 17] | 3.53 [2.47 to 5.06]
  B (Day 22 / Day1) | 12 [7.69 to 18] | 2.51 [1.93 to 3.27]

4. Primary Outcome: Percentages of Subjects With HI Titer ≥40 After 1 Dose of Cell Culture Derived Vaccine (cTIV).
Description: HI titer as assessed by hemagglutination inhibition (HI) assay using egg derived antigen in adults and elderly subjects.
  This criterion is met according to European (CHMP) guideline if the percentages of subjects achieving HI titers ≥40 is >70% for adults and >60% for elderly subjects.
Time Frame: 3 weeks postvaccination (Day 22)
Population: Analysis was done on per protocol set
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | cTIV (Adults) | cTIV (Elderly)
Number analyzed (Participants) | 68 | 67
Percentages of Subjects
  A/H1N1 Prevaccination (Day 1) | 35 [24 to 48] | 37 [26 to 50]
  A/H1N1 Postvaccination (Day 22) | 96 [88 to 99] | 96 [87 to 99]
  A/H3N2 Prevaccination (Day 1) | 51 [39 to 64] | 72 [59 to 82]
  A/H3N2 Postvaccination (Day 22) | 97 [90 to 100] | 96 [87 to 99]
  B Prevaccination (Day 1) | 13 [6 to 24] | 28 [18 to 41]
  B Postvaccination (Day 22) | 79 [68 to 88] | 66 [53 to 77]

5. Primary Outcome: Percentages of Subjects With Seroconversion or Significant Increase After 1 Dose of Cell Culture Derived Vaccine (cTIV).
Description: Proportion of subjects with either seroconversion (antibody increase from < 10 pre vaccination to ≥40 post vaccination) or significant increase (antibody titer of ≥10 pre vaccination and 4-fold antibody increase post vaccination).
  According to the CHMP criteria, the percentages of subjects achieving seroconversion or significant increase should be >40% for adults and >30% for elderly subjects.
Time Frame: 3 weeks postvaccination (Day 22)
Population: Analysis was done on per protocol set
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | cTIV (Adults) | cTIV (Elderly)
Number analyzed (Participants) | 68 | 67
Percentages of Subjects
  A/H1N1 | 79 [68 to 88] | 67 [55 to 78]
  A/H3N2 | 72 [60 to 82] | 40 [28 to 53]
  B | 65 [52 to 76] | 25 [16 to 37]

ADVERSE EVENTS:
Time Frame: All solicited adverse reactions were collected from Day 0 - Day 3. All unsolicited adverse events and Serious adverse events were collected throughout study period (Day 0- Day 21).
Arm/Group | cTIV (Adults) | cTIV (Elderly)
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/67
Other Adverse Events (participants affected / at risk) | 40/68 | 21/67
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | cTIV (Adults) (N=68) | cTIV (Elderly) (N=67)
Fatigue (General disorders) | 10 | 8
Injection site induration (General disorders) | 5 | 5
Injection site pain (General disorders) | 31 | 16
Malaise (General disorders) | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Headache (Nervous system disorders) | 12 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days